CLINICAL TRIAL: NCT00223119
Title: Comparison of Absorbable Sutures in Perineal Laceration Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study recruitment very slow.
Sponsor: Medtronic - MITG (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SYN03001
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Perineal Laceration Repair
Keywords: perineal trauma; perineal laceration; persistent perineal pain

INTERVENTIONS:
Device: Absorbable Sutures

SUMMARY:
The purpose of this study is to determine the difference in pain scales between absorbable suture types for second-degree perineal laceration repair.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to sign informed consent
* Vaginal laceration that requires sutures but does not involve the anal sphincter (third-degree tear) or rectal mucosa (fourth-degree tear)

Exclusion Criteria:

* Inability to speak and understand English or Spanish
* Previous diagnosis of vulvodynia, dyspareunia, or other chronic vulvar pain syndrome
* Extensive perineal warts or vulvar varicosities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Doran, Study Director — Medtronic - MITG
Locations (1):
- US Surgical, Norwalk, Connecticut, United States